CLINICAL TRIAL: NCT03969901
Title: A Phase 2/3 Open-label, Randomized, Active-controlled Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of MK-7655A in Pediatric Participants From Birth to Less Than 18 Years of Age With Confirmed or Suspected Gram-negative Bacterial Infection
Brief Title: Safety, Tolerability, Efficacy and Pharmacokinetics of Imipenem/Cilastatin/Relebactam (MK-7655A) in Pediatric Participants With Gram-negative Bacterial Infection (MK-7655A-021)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7655A-021; MK-7655A-021 (Other: MSD); 2019-000338-20 (EudraCT Number)
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Suspected or Documented Gram-negative Bacterial Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMI/REL (Experimental): Participants with cIAI or cUTI will receive imipenem/cilastatin/relebactam (IMI/REL) via IV infusion for a minimum of 5 days (with optional investigator's choice of locally sourced oral switch medication after 3 days) up to a maximum of 14 days. Participants with HABP/VABP will receive IMI/REL via IV infusion for a minimum of 7 days up to a maximum of 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection will receive IMI/REL via IV infusion for 14 days. All oral switch medications will be chosen from a list of acceptable approved agents and will be administered per authorized Package Insert (PI), Summary of Product Characteristics (SPC), or international treatment guidelines.
  Interventions: Drug: IMI/REL; Drug: Oral Switch
- Active Control (Active Comparator): Participants with cIAI or cUTI will receive active control via IV infusion for a minimum of 5 days (with optional investigator's choice of locally sourced oral switch medication after 3 days) up to a maximum of 14 days. Participants with HABP/VABP will receive active control via IV infusion for a minimum of 7 days up to a maximum of 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection will receive active control via IV infusion for 14 days. All active control and oral switch medications will be administered per authorized PI, SPC, or international treatment guidelines. All active control and oral switch medications will be chosen from a list of acceptable approved agents.
  Interventions: Drug: Active Control; Drug: Oral Switch

INTERVENTIONS:
Drug: IMI/REL — Age-based dosing:
  * 12 to <18 years, IMI 500 and REL 250 mg, IV infusion every 6 hours
  * 6 to <12 years, IMI 15 and REL 7.5 mg/kg, IV infusion every 6 hours
  * 2 to <6 years, IMI 15 and REL 7.5 mg/kg, IV infusion every 6 hours
  * 3 months to <2 years, IMI 15 and REL 7.5 mg/kg, IV infusion every 6 hours
  * Birth to <3 months, IMI 15 and REL 7.5 mg/kg, IV infusion every 8 hours NOTE: Participants with cIAI or cUTI may be switched to oral therapy after at least 3 days of IV study intervention.
  Other Names: MK-7655A
  Arms: IMI/REL
Drug: Active Control — All active control medications will be chosen from a list of acceptable approved agents for each infection type (HABP or VABP, cIAI, and UTI) and will be given via IV infusion, per authorized Package Insert (PI), Summary of Product Characteristics (SPC), or international treatment guidelines.
  NOTE: Participants with cIAI or cUTI may be switched to oral therapy after at least 3 days of IV study intervention. All oral switch medications will be chosen from a list of acceptable approved agents.
  Arms: Active Control
Drug: Oral Switch — All oral switch medications will be investigator's choice from a list of acceptable approved agents for infection types cIAI, and cUTI and will be given per authorized Package Insert (PI), Summary of Product Characteristics (SPC), or international treatment guidelines. Participants with cIAI or cUTI may be switched to oral therapy after at least 3 days of IV study intervention.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of imipenem/cilastatin/relebactam (IMI/REL) in participants from birth to less than 18 years of age with confirmed or suspected gram-negative bacterial infection. Participants are expected to require hospitalization through completion of intravenous (IV) study intervention, and have at least one of the following primary infection types: hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP); complicated intra-abdominal infection (cIAI); or complicated urinary tract infection (cUTI). Participants will be randomized in a 3:1 ratio to receive IMI/REL or active control. This study will also evaluate the efficacy of IMI/REL by assessing all-cause mortality at Day 28 post-randomization, as well as clinical and microbiological response to treatment. It will also evaluate the pharmacokinetics of IMI/REL.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include but are not limited to:

* Requires hospitalization and treatment with intravenous (IV) antibacterial therapy for confirmed or suspected gram-negative bacterial infection (in the absence of meningitis), and is expected to require hospitalization through completion of IV study intervention, with at least 1 of the following primary infection types: Hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP); complicated intra-abdominal infection (cIAI); or complicated urinary tract infection (cUTI).
* For Age Cohorts 4 and 5, participant is at least 37 weeks postmenstrual age at the time of signing the informed consent/assent.
* If female, must not be pregnant or breastfeeding, and at least 1 of the following conditions must apply: must not be a woman of childbearing potential (WOCBP); OR, if a WOCBP, must agree to follow contraceptive guidance during the intervention period and for at least 24 hours after the last dose of study intervention.
* Has sufficient intravascular access to receive study drug through an existing peripheral or central line.

Exclusion Criteria:

Exclusion Criteria include but are not limited to:

* Is expected to survive less than 72 hours.
* Has a concurrent infection that would interfere with evaluation of response to the study antibacterials (imipenem/cilastatin/relebactam (IMI/REL) or Active Control), including any of the following: endocarditis; osteomyelitis; meningitis; prosthetic joint infection; active pulmonary tuberculosis; disseminated fungal infection; concomitant infection at the time of randomization that requires non-study systemic antibacterial therapy in addition to IV study treatment or oral step-down therapy (medications with only gram-positive activity [e.g., vancomycin, linezolid] are allowed).
* Has HABP/VABP caused by an obstructive process, including lung cancer (or other malignancy metastatic to the lungs resulting in pulmonary obstruction) or other known obstruction.
* Has a cUTI, with any of the following: complete obstruction of any portion of the urinary tract (i.e., requiring a permanent indwelling urinary catheter or instrumentation); documented reflux of ileal loop urinary diversion; suspected or confirmed perinephric or intrarenal abscess; suspected or confirmed prostatitis, urethritis, or epididymitis; trauma to pelvis/urinary tract; presence of indwelling urinary catheter which cannot be removed at study entry.
* Has any of the following medical conditions at screening: history of a seizure disorder (requiring ongoing treatment with anti-convulsive therapy or prior treatment with anti-convulsive therapy within the last 3 years); cystic fibrosis; history of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to IMI, or to any carbapenem, cephalosporin, penicillin, or other β-lactam agent, or to other β-lactamase inhibitors (e.g., tazobactam, sulbactam, clavulanic acid, avibactam).
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might expose the participant to risk by participating in the study, confound study results, or interfere with the participant's participation for the full duration of the study.
* If less than 3 months of age, has received more than 72 hours of empiric antibacterial treatment for suspected meningitis prior to initiation of IV study intervention.
* For all Age Cohorts, provided all other eligibility criteria are met, the following participants may be enrolled:

  * A participant failing prior antibiotic therapy for a current episode of cUTI or HABP/VABP who: Has received the prior antibacterial treatment for at least 48 hours; Has persistent clinical or radiographic findings clearly indicating ongoing infection; Fulfills other laboratory or microbiology criteria for enrollment
  * A participant failing prior antibiotic therapy for a current episode of cIAI who: Has received the prior antibacterial treatment for at least 48 hours; Has persistent clinical or radiographic findings clearly indicating ongoing infection; Fulfills other laboratory or microbiology criteria for enrollment; Has planned operative intervention no more than 24 hours after first dose of study treatment; Has not received any further nonstudy antibiotics postoperatively
* If 3 months of age or older, or <3 months of age without suspected meningitis, has received potentially therapeutic antibacterial therapy (e.g., with gram-negative activity), including bladder infusions with topical urinary antiseptics or antibacterial agents, for a duration of more than 24 hours during the 48 hours preceding the first dose of study intervention.
* Is anticipated to be treated with any of the following medications: valproic acid or divalproex sodium (or has used valproic acid or divalproex sodium in the 2 weeks prior to screening) through 24 hours after completion of the final dose of IV study intervention for participants who receive IMI/REL or carbapenem; concomitant IV, oral, or inhaled antimicrobial agents with gram-negative activity, in addition to those designated in the study intervention groups, during the course of all (IV/oral) study intervention; planned receipt of suppressive/prophylactic antibiotics with gram-negative activity after completion of study intervention.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 30 days prior to screening.
* Has enrolled previously in the current study and been discontinued or has received REL for any other reason.
* Has an estimated creatinine clearance (based on the Cockcroft-Gault equation, for participants ≥12 years of age or estimated glomerular filtration rate (eGFR), based on the modified Schwartz equation, for participants <12 years of age below that specified for the appropriate age range; or requires peritoneal dialysis, hemodialysis, or hemofiltration.
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥5 × upper limit of normal (ULN) at the time of screening. NOTE: Patients with acute hepatic failure or acute decompensation of chronic hepatic failure should also be excluded.
* Is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (67):
- United States (8):
  - Banner University Medical Center ( Site 0356), Tucson, Arizona
  - Miller Children's & Women's Hospital ( Site 0349), Long Beach, California
  - Rady Children's Hospital-San Diego ( Site 0347), San Diego, California
  - Tufts Medical Center-Floating Hospital for Children ( Site 0350), Boston, Massachusetts
  - University of New Mexico ( Site 0358), Albuquerque, New Mexico
  - University Hospital ( Site 0360), San Antonio, Texas
  - Children's Hospital of Richmond at VCU ( Site 0359), Richmond, Virginia
  - West Virginia University Ruby Memorial Hospital ( Site 0344), Morgantown, West Virginia
- Bulgaria (6):
  - UMHAT Deva Maria. EOOD ( Site 0165), Burgas
  - MHAT City Clinic Sv. Georgi EOOD ( Site 0167), Montana
  - UMHAT Dr. Georgi Stranski EAD ( Site 0174), Pleven
  - UMHAT Kanev AD ( Site 0168), Rousse
  - UMHAT Kanev AD ( Site 0169), Rousse
  - MHAT Dr. Ival Seliminski ( Site 0173), Sliven
- Hospital Roberto del Río ( Site 0802), Santiago, Region M. de Santiago, Chile
- Colombia (5):
  - Fundacion Hospital San Vicente de Paul ( Site 0269), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0264), Barranquilla, Atlántico
  - Sociedad de Cirugía de Bogotá - Hospital de San Jose ( Site 0265), Bogotá, Bogota D.C.
  - Fundacion Hospital Infantil Universitario de San Jose ( Site 0268), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 0266), Cali, Valle del Cauca Department
- Tallinn Children Hospital ( Site 0209), Tallinn, Harju, Estonia
- France (3):
  - Hopitaux Pediatriques CHU Lenval ( Site 0143), Nice, Alpes-Maritimes
  - Hopital Francois Mitterand ( Site 0146), Dijon, Cote-d Or
  - Hopital Jeanne de Flandre ( Site 0145), Lille, Hauts-de-France
- Greece (3):
  - University of Athens - Aghia Sophia Childrens Hospital ( Site 0243), Athens, Attica
  - Pan and Aglaia Kyriakou Children s Hospital ( Site 0247), Athens, Attica
  - Hippokration General Hospital of Thessaloniki ( Site 0244), Thessaloniki
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont ( Site 0100), Debrecen, Hajdú-Bihar
  - Szabolcs-Szatmar-Bereg Megyei Kórházak és Egyetemi Otatókórház-Gyermekosztály ( Site 0105), Nyíregyháza, Szabolcs-Szatmár-Bereg
- Israel (4):
  - Rambam Medical Center ( Site 0189), Haifa
  - Hadassah Ein Karem Hebrew University Medical Center ( Site 0188), Jerusalem
  - Schneider Children's Medical Center ( Site 0187), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0190), Ramat Gan
- Mexico (4):
  - Hospital General de Tijuana ( Site 0284), Tijuana, Estado de Baja California
  - Hospital del Nino y Adolescente Morelense ( Site 0286), Emiliano Zapata, Morelos
  - Centenario Hospital Miguel Hidalgo-Pediatrics Department ( Site 0290), Aguascalientes
  - Instituto Nacional de Pediatria ( Site 0291), Mexico City
- Haukeland Universitetssjukehus ( Site 0500), Bergen, Hordaland, Norway
- Philippines (2):
  - University of the Philippines-Philippine General Hospital ( Site 0318), Manila, National Capital Region
  - Philippine Children s Medical Center ( Site 0317), Quezon City, National Capital Region
- Poland (3):
  - Wojewodzki Szpital Zespolony im. Rydgiera ( Site 0220), Torun, Kuyavian-Pomeranian Voivodeship
  - SPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 0226), Łomianki, Masovian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki ( Site 0223), Lodz, Łódź Voivodeship
- Russia (8):
  - Pediatric Hematology Oncology and Immunology Centre n.a. D.Rogachev. ( Site 0233), Moscow, Moscow
  - Morozovskaya Children City Clinical Hospital ( Site 0241), Moscow, Moscow
  - State Budgetary Healthcare Institution of Novosibirsk Region City Childrens Clinical Emergency Hospi, Novosibirsk, Novosibirsk Oblast
  - Children s City Clinical Hospital 5 n.a. N.F. Filatov ( Site 0235), Saint Petersburg, Sankt-Peterburg
  - St.Petersburg State Pediatric Medical University ( Site 0236), Saint Petersburg, Sankt-Peterburg
  - Children's City Clinical Hospital #1 ( Site 0237), Saint Petersburg, Sankt-Peterburg
  - Smolensk Regional Clinical Hospital ( Site 0231), Smolensk, Smolensk Oblast
  - Regional Childrens Clinical Hospital ( Site 0400), Vologda, Vologda Oblast
- South Africa (3):
  - Empilweni Services and Research Unit ( Site 1557), Johannesburg, Gauteng
  - Chris Hani Baragwanath Academic Hospital ( Site 0156), Johannesburg, Gauteng
  - Molotlegi Street ( Site 0155), Pretoria, Gauteng
- Spain (3):
  - Hospital Infantil Universitario Nino Jesus ( Site 0114), Madrid
  - Hospital Universitario La Paz ( Site 0113), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 0115), Seville
- Turkey (Türkiye) (5):
  - Cukurova University Medical Faculty ( Site 0200), Adana
  - Ankara Universitesi Tip Fakultesi. ( Site 0202), Ankara
  - Eskisehir Osmangazi University Medical ( Site 0201), Eskişehir
  - SBU Sariyer Hamidiye Etfal Egitim ve Arastirma Hastanesi ( Site 0198), Istanbul
  - Ege Universitesi Tıp Fakultesi Hastanesi ( Site 0199), Izmir
- Ukraine (5):
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 0121), Dnipro, Dnipropetrovsk Oblast
  - Communal non-commercial enterprise "Kryvorizka city clinical hospital 16" of Kryvyy Rig city council, Kryvyy Rig, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Children Clinical Hospital ( Site 0131), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kharkiv City Children Hospital 16 ( Site 0130), Kharkiv, Kharkivs’ka Oblast’
  - Municipal Enterprise Children's City Clinical Hospital in Poltava City Council ( Site 0122), Poltava, Poltava Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26857&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- IMI/REL Age Cohort 1: Adolescents (12 to <18 Years): Participants with cIAI and complicated urinary tract infection cUTI received IMI/REL fixed-dose combination of 500 mg/250 mg via IV infusion every 6 hours for a minimum of 5 days with an option of investigator's choice of locally sourced oral switch medication after a minimum of 3 days of IV therapy alone. Participants with HABP/VABP received IMI/REL fixed-dose combination of 500 mg/250 mg via IV infusion every 6 hours for 7 days up to 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received IMI/REL fixed-dose combination of 500 mg/250 mg via IV infusion every 6 hours for 14 days. All oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All oral switch medications were chosen from a list of acceptable approved agents.
- Active Control Age Cohort 1: Adolescents (12 to <18 Years); Active Control Age Cohort 2: Older Children (6 to <12 Years); Active Control Age Cohort 3: Younger Children (2 to <6 Years); Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years); Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months): Participants with cIAI or cUTI received investigator's choice of locally sourced active control via IV infusion for a minimum of 5 days (with optional investigator's choice of locally sourced oral switch medication after 3 days of IV therapy alone) up to a maximum of 14 days. Participants with HABP/VABP received investigator's choice of locally sourced active control via IV infusion for a minimum of 7 days up to a maximum of 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received investigator's choice of locally sourced active control via IV infusion for 14 days. All active control and oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All active control and oral switch medications were chosen from a list of acceptable approved agents.
- IMI/REL Age Cohort 2: Older Children (6 to <12 Years); IMI/REL Age Cohort 3: Younge Children (2 to <6 Years); IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years): Participants with cIAI and cUTI received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 6 hours for a minimum of 5 days with an option of investigator's choice of locally sourced oral switch medication after a minimum of 3 days of IV therapy alone. Participants with HABP/VABP received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 6 hours for 7 days up to 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 6 hours for 14 days. All oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All oral switch medications were chosen from a list of acceptable approved agents.
- IMI/REL Age Cohort 5 Neonates and Young Infants (Birth to <3 Months): Participants with cIAI and cUTI received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 8 hours for a minimum of 5 days with an option of investigator's choice of locally sourced oral switch medication after a minimum of 3 days of IV therapy alone. Participants with HABP/VABP received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 8 hours for 7 days up to 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 8 hours for 14 days. All oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All oral switch medications were chosen from a list of acceptable approved agents.
Period: Overall Study
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younge Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5 Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Started | 10 | 2 | 31 | 11 | 22 | 8 | 15 | 5 | 8 | 3
Treated | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Completed | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- IMI/REL Age Cohort 3: Younger Children (2 to <6 Years); IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years): Participants with cIAI and cUTI received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 6 hours for a minimum of 5 days with an option of investigator's choice of locally sourced oral switch medication after a minimum of 3 days of IV therapy alone. Participants with HABP/VABP received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 6 hours for 7 days up to 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 6 hours for 14 days. All oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All oral switch medications were chosen from a list of acceptable approved agents.
- IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months): Participants with cIAI and cUTI received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 8 hours for a minimum of 5 days with an option of investigator's choice of locally sourced oral switch medication after a minimum of 3 days of IV therapy alone. Participants with HABP/VABP received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 8 hours for 7 days up to 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received IMI/REL fixed-dose combination of 15 mg/7.5 mg via IV infusion every 8 hours for 14 days. All oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All oral switch medications were chosen from a list of acceptable approved agents.
- Total: Total of all reporting groups
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Total
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 22 | 8 | 15 | 5 | 8 | 3 | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.1 (2.0) | 16.5 (0.7) | 8.4 (1.7) | 8.0 (1.7) | 3.5 (1.1) | 4.3 (1.2) | 0.9 (0.5) | 0.7 (0.6) | 0.1 (0.1) | 0.1 (0.1) | 5.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 13 | 8 | 12 | 3 | 7 | 1 | 3 | 0 | 56
  Male | 2 | 1 | 18 | 3 | 10 | 5 | 8 | 4 | 5 | 3 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 9 | 1 | 12 | 4 | 5 | 1 | 3 | 2 | 43
  Not Hispanic or Latino | 5 | 1 | 21 | 10 | 10 | 4 | 9 | 4 | 5 | 1 | 70
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  White | 7 | 1 | 27 | 10 | 19 | 4 | 11 | 5 | 8 | 2 | 94
  More than one race | 3 | 1 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection Type [Count of Participants; unit: Participants] — Infection type for this study indicates one of three types of infections: complicated intraabdominal infection (cIAI); complicated urinary tract infection (cUTI); or hospital acquired bacterial pneumonia/ventilator acquired bacterial pneumonia (HABP/VABP)
  Participants
    cIAI | 5 | 1 | 21 | 7 | 14 | 5 | 0 | 1 | 0.0 | 0.0 | 54
    cUTI | 4 | 1 | 10 | 4 | 6 | 2 | 14 | 4 | 7 | 3 | 55
    HABP/VABP | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with AEs are presented.
Time Frame: Up to 28 days
Population: All randomized participants who received at least 1 dose of IV study intervention. Participants were included in the treatment group to which they were randomized.
Measure: Number; unit: Percentage of Participants
Groups:
- Active Control Cohort 1: Adolescents: (12 to <18 Years); Active Control Age Cohort 2: Older Children (6 to <12 Years); Active Control Age Cohort 3: Younger Children (2 to <6 Years); Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years); Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months): Participants with cIAI or cUTI received investigator's choice of locally sourced active control via IV infusion for a minimum of 5 days (with optional investigator's choice of locally sourced oral switch medication after 3 days of IV therapy alone) up to a maximum of 14 days. Participants with HABP/VABP received investigator's choice of locally sourced active control via IV infusion for a minimum of 7 days up to a maximum of 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received investigator's choice of locally sourced active control via IV infusion for 14 days. All active control and oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All active control and oral switch medications were chosen from a list of acceptable approved agents.
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Cohort 1: Adolescents: (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Percentage of Participants | 60.0 | 50.0 | 64.5 | 36.4 | 71.4 | 62.5 | 93.3 | 50.0 | 25.0 | 66.7

2. Primary Outcome: Percentage of Participants Who Discontinued Study Medication Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study medication due to an AE are presented.
Time Frame: Up to 14 days
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Cohort 1: Adolescents: (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Percentage of Participants | 0.0 | 0.0 | 12.9 | 9.1 | 0.0 | 0.0 | 6.7 | 25.0 | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants With All-cause Mortality Through Day 28
Description: For each participant, survival status was assessed at Day 28 post-randomization. The percentage of participants with all-cause mortality through Day 28 is presented.
Time Frame: Up to Day 28
Population: The analysis population included all randomized participants who received at least 1 dose of IV study intervention. Participants were included in the treatment group to which they were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at End of Therapy (EOT)
Description: A favorable clinical response at EOT requires an assessment of "cure" or "improved". Cure is defined as all preintervention signs and symptoms of the index infection have resolved (or returned to "preinfection status", with no new symptoms) AND no additional antibacterial intervention is required for the index infection. Improved is defined as the majority of preintervention signs and symptoms of the index infection have improved or resolved (or returned to "preinfection status", with no new symptoms) AND no additional antibacterial intervention is required. The percentage of participants with a favorable clinical response at EOT is presented.
Time Frame: Day 5 up to Day 14
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Active Control Age Cohort 1: Adolescents (12 to 18 Years); Active Control Age Cohort 2: Older Children (6 to <12 Years); Active Control Age Cohort 3: Younger Children (2 to <6 Years); Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years); Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months): Participants with cIAI or cUTI received investigator's choice of locally sourced active control via IV infusion for a minimum of 5 days (with optional investigator's choice of locally sourced oral switch medication after 3 days of IV therapy alone) up to a maximum of 14 days. Participants with HABP/VABP received investigator's choice of locally sourced active control via IV infusion for a minimum of 7 days up to a maximum of 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received investigator's choice of locally sourced active control via IV infusion for 14 days. All active control and oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All active control and oral switch medications were chosen from a list of acceptable approved agents.
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to 18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Percentage of Participants | 90.0 [57.4 to 100.0] | 50.0 [9.5 to 90.5] | 77.4 [59.9 to 88.9] | 81.8 [51.2 to 96.0] | 90.5 [69.9 to 98.6] | 87.5 [50.8 to 99.9] | 53.3 [30.1 to 75.2] | 75.0 [28.9 to 96.6] | 87.5 [50.8 to 99.9] | 33.3 [5.6 to 79.8]

5. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Early Follow-Up (EFU)
Description: A favorable clinical response at EFU requires an assessment of "cure" or "sustained cure". Cure is defined as all preintervention signs and symptoms of the index infection have resolved (or returned to "preinfection status", with no new symptoms) AND no additional antibacterial intervention is required for the index infection. Sustained cure is defined as a clinical response for the prior visit (EOT or EFU) being defined as "cure". The percentage of participants with a favorable clinical response at EFU is presented.
Time Frame: Day 12 up to Day 28
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Percentage of Participants | 90.0 [57.4 to 100.0] | 50.0 [9.5 to 90.5] | 77.4 [59.9 to 88.9] | 81.8 [51.2 to 96.0] | 85.7 [64.5 to 95.9] | 87.5 [50.8 to 99.9] | 26.7 [10.5 to 52.4] | 75.0 [28.9 to 96.6] | 62.5 [30.4 to 86.5] | 33.3 [5.6 to 79.8]

6. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Late Follow-Up (LFU)
Description: A favorable clinical response at LFU requires an assessment of "cure" or "sustained cure". Cure is defined as all preintervention signs and symptoms of the index infection have resolved (or returned to "preinfection status", with no new symptoms) AND no additional antibacterial intervention is required for the index infection. Sustained cure is defined as a clinical response for the prior visit (EOT or EFU) being defined as "cure". The percentage of participants with a favorable clinical response at LFU is presented.
Time Frame: Baseline and Day 19 up to Day 42
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 2 | 31 | 11 | 21 | 8 | 15 | 4 | 8 | 3
Percentage of Participants | 90.0 [57.4 to 100.0] | 50.0 [9.5 to 90.5] | 74.2 [56.5 to 86.5] | 81.8 [51.2 to 96.0] | 81.0 [59.4 to 92.9] | 87.5 [50.8 to 99.9] | 33.3 [15.0 to 58.5] | 75.0 [28.9 to 96.6] | 62.5 [30.4 to 86.5] | 33.3 [5.6 to 79.8]

7. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at End of Therapy (EOT)
Description: A favorable microbial response is defined as eradication or presumed eradication. Eradication is defined as one of the following: A lower respiratory tract culture taken at the EOT visit shows eradication of the pathogen found at study entry for HABP/VABP; An intra-abdominal culture taken at the EOT visit shows eradication of the pathogen found at study entry for cIAI; A urine culture taken at the EOT visit shows eradication of the uropathogen (reduced to <103 CFU/mL) found at study entry for cUTI. Presumed eradication is defined as no specimen taken because participant is deemed clinically improved or cured of the pathogen found at study entry. The percentage of participants with a favorable microbial response at EOT is presented.
Time Frame: Day 5 up to Day 14
Population: For participants with HABP/VABP and cIAI: Has received at least 1 dose of IV study intervention; AND baseline infection-site culture grew at least 1 gram-negative pathogenic organism. For participants with cUTI: Has received at least 1 dose of IV study intervention; AND baseline urine culture grew at least 1 gram-negative pathogenic organism at sufficient quantity (ie, growth at ≥105 CFU/mL of uropathogen). Participants were included in the intervention group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 7 | 1 | 27 | 10 | 16 | 5 | 11 | 4 | 7 | 2
Percentage of Participants | 100.0 [59.6 to 100.0] | 100.0 [16.7 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [67.9 to 100.0] | 100.0 [77.3 to 100.0] | 100.0 [51.1 to 100.0] | 72.7 [42.9 to 90.8] | 75.0 [28.9 to 96.6] | 100.0 [59.6 to 100.0] | 50.0 [9.5 to 90.5]

8. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at End of Follow-Up (EFU)
Description: A favorable microbiological response at EFU is defined as eradication or presumed eradication. Eradication is defined as one of the following: A lower respiratory tract culture taken at the EFU visit shows eradication of the pathogen found at study entry for HABP/VABP; An intra-abdominal culture taken at the EFU visit shows eradication of the pathogen found at study entry for cIAI; A urine culture taken at the EFU visit shows eradication of the uropathogen (reduced to <103 CFU/mL) found at study entry for cUTI. Presumed eradication is defined as no specimen taken because participant is deemed clinically improved or cured of the pathogen found at study entry. The percentage of participants with a favorable microbial response at EFU is presented.
Time Frame: Day 12 up to Day 28
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 7 | 1 | 27 | 10 | 16 | 5 | 11 | 4 | 7 | 2
Percentage of Participants | 71.4 [35.2 to 92.4] | 100.0 [16.7 to 100.0] | 96.3 [80.2 to 100.0] | 100.0 [67.9 to 100.0] | 93.8 [69.7 to 100.0] | 100.0 [51.1 to 100.0] | 63.6 [35.2 to 85.0] | 75.0 [28.9 to 96.6] | 71.4 [35.2 to 92.4] | 50.0 [9.5 to 90.5]

9. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Late Follow-Up (LFU)
Description: A favorable microbiological response at LFU is defined as eradication or presumed eradication. Eradication is defined as one of the following: A lower respiratory tract culture taken at the LFU visit shows eradication of the pathogen found at study entry for HABP/VABP; An intra-abdominal culture taken at the LFU visit shows eradication of the pathogen found at study entry for cIAI; A urine culture taken at the LFU visit shows eradication of the uropathogen (reduced to <103 CFU/mL) found at study entry for cUTI. Presumed eradication is defined as no specimen taken because participant is deemed clinically improved or cured of the pathogen found at study entry. The percentage of participants with a favorable microbial response at LFU is presented.
Time Frame: Day 19 up to Day 42
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 7 | 1 | 27 | 10 | 16 | 5 | 11 | 4 | 7 | 2
Percentage of Participants | 85.7 [46.7 to 99.5] | 0.0 [0.0 to 83.3] | 96.3 [80.2 to 100.0] | 100.0 [67.9 to 100.0] | 87.5 [62.7 to 97.8] | 100.0 [51.1 to 100.0] | 72.7 [42.9 to 90.8] | 75.0 [28.9 to 96.6] | 71.4 [35.2 to 92.4] | 50.0 [9.5 to 90.5]

10. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours (AUC0-24) of Imipenem Following Administration of IMI/REL
Description: AUC0-24 is a measure of the total amount of drug in the plasma from the dose to Hour 24. Blood samples were collected to determine the AUC0-24 of imipenem.
Time Frame: On Day 1 at 30 minutes prior to start of first IV infusion of study drug, at end of first infusion, and 2 to 6 hours after start of first infusion; and once at on-therapy visit (Day 2 or Day 3) at 2 to 6 hours after start of any infusion that day.
Population: The analysis population includes all participants who received at least 1 dose of IMI/REL and had at least one measurable pharmacokinetic (PK) sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Groups:
- IMI/REL Age Cohort 1: Adolescents: (12 to <18 Years): Participants with cIAI and complicated urinary tract infection cUTI received IMI/REL fixed-dose combination of 500 mg/250 mg via IV infusion every 6 hours for a minimum of 5 days with an option of investigator's choice of locally sourced oral switch medication after a minimum of 3 days of IV therapy alone. Participants with HABP/VABP received IMI/REL fixed-dose combination of 500 mg/250 mg via IV infusion every 6 hours for 7 days up to 14 days. Participants with bacteremia or Pseudomonas aeruginosa infection received IMI/REL fixed-dose combination of 500 mg/250 mg via IV infusion every 6 hours for 14 days. All oral switch medications were administered per authorized PI, SPC, or international treatment guidelines. All oral switch medications were chosen from a list of acceptable approved agents.
Arm/Group | IMI/REL Age Cohort 1: Adolescents: (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 31 | 21 | 15 | 8
µM*hr | 610 (55.5) | 720 (25.8) | 692 (23.5) | 788 (28.4) | 795 (19.5)

11. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours (AUC0-24) of Relebactam Following Administration of IMI/REL
Description: AUC0-24 is a measure of the total amount of drug in the plasma from the dose to Hour 24. Blood samples were collected to determine the AUC0-24 of relebactam.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 31 | 21 | 15 | 8
µM*hr | 399 (64) | 469 (30.9) | 459 (30.4) | 634 (56.8) | 605 (50.1)

12. Secondary Outcome: Concentration at End of Infusion (Ceoi) of Imipenem Following Administration of IMI/REL
Description: Ceoi is the concentration of the drug at the end of infusion. Blood samples for analysis were collected within 10 minutes of the end of infusion to determine the Ceoi of imipenem.
Time Frame: At the end of the first infusion on Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 31 | 21 | 15 | 8
µM | 79.2 (17.6) | 103 (15) | 101 (12.7) | 109 (14.1) | 117 (5.51)

13. Secondary Outcome: Concentration at End of Infusion (Ceoi) of Relebactam Following Administration of IMI/REL
Description: Ceoi is the concentration of the drug at the end of infusion. Blood samples for analysis were collected within 10 minutes of the end of infusion to determine the Ceoi of relebactam.
Time Frame: At the end of the first infusion on Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 10 | 31 | 21 | 15 | 8
µM | 43.4 (28.6) | 56.1 (18.6) | 56.1 (16.2) | 67.1 (27.4) | 67.9 (22.2)

14. Secondary Outcome: Percentage of Time Imipenem Concentration Is Above Minimum Inhibitory Concentration (%T>MIC of Imipenem) Following Administration of IMI/REL
Description: Percentage of Time Imipenem Concentration Is Above Minimum Inhibitory Concentration (%T>MIC) is defined as the cumulative percentage the drug concentration exceeds the MIC at steady state pharmacokinetic conditions. Blood samples were collected to determine %T>MIC of imipenem. %T>MIC is calculated using baseline microbiological response values.
Time Frame: as for outcome 10
Population: The analysis population includes all participants who received at least 1 dose of IMI/REL and had at least one measurable pharmacokinetic (PK) sample for %T>MIC.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
Number analyzed (Participants) | 6 | 22 | 15 | 8 | 6
Percentage of time | 100.0 (0.0) | 93.4 (22.1) | 83.6 (23.1) | 79.6 (35.3) | 83.5 (25.6)

ADVERSE EVENTS:
Time Frame: Up to 42 days
Description: All-cause mortality: all randomized participants; Safety: all randomized participants who received at least one dose of study treatment.
Arm/Group | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) | Active Control Age Cohort 2: Older Children (6 to <12 Years) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/31 | 0/11 | 0/22 | 0/8 | 0/15 | 0/5 | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 6/31 | 1/11 | 0/21 | 0/8 | 4/15 | 1/4 | 0/8 | 1/3
Other Adverse Events (participants affected / at risk) | 6/10 | 1/2 | 17/31 | 3/11 | 13/21 | 5/8 | 12/15 | 2/4 | 2/8 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) (N=10) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) (N=2) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) (N=31) | Active Control Age Cohort 2: Older Children (6 to <12 Years) (N=11) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) (N=21) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) (N=8) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) (N=15) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) (N=4) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) (N=8) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) (N=3)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMI/REL Age Cohort 1: Adolescents (12 to <18 Years) (N=10) | Active Control Age Cohort 1: Adolescents (12 to <18 Years) (N=2) | IMI/REL Age Cohort 2: Older Children (6 to <12 Years) (N=31) | Active Control Age Cohort 2: Older Children (6 to <12 Years) (N=11) | IMI/REL Age Cohort 3: Younger Children (2 to <6 Years) (N=21) | Active Control Age Cohort 3: Younger Children (2 to <6 Years) (N=8) | IMI/REL Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) (N=15) | Active Control Age Cohort 4: Infants and Toddlers (3 Months to <2 Years) (N=4) | IMI/REL Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) (N=8) | Active Control Age Cohort 5: Neonates and Young Infants (Birth to <3 Months) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 5 (15) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 4 (5) | 3 (5) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine urine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pH urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urethral fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03969901/Prot_SAP_000.pdf